CLINICAL TRIAL: NCT00429299
Title: Chemotherapy Plus Lapatinib or Trastuzumab or Both in Her2+ Primary Breast Cancer. A Randomized Phase IIb Study With Biomarker Evaluation.
Brief Title: Neoadjuvant Study With Chemotherapy, Lapatinib And Trastuzumab In Breast Cancer
Acronym: CHERLOB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGF106988
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-01

CONDITIONS: Neoplasms, Breast
Keywords: neo-adjuvant trastuzumab early breast cancer lapatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Trastuzumab; Paclitaxel; Fluorouracil; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Active Comparator): Chemotherapy plus trastuzumab
  Interventions: Biological: trastuzumab; Drug: paclitaxel; Drug: fluorouracil; Drug: epidoxorubicin; Drug: cyclophosphamide
- Arm B (Experimental): Chemotherapy plus lapatinib
  Interventions: Drug: lapatinib; Drug: paclitaxel; Drug: fluorouracil; Drug: epidoxorubicin; Drug: cyclophosphamide
- Arm C (Active Comparator): Chemotherapy plus trastuzumab plus lapatinib
  Interventions: Drug: lapatinib; Biological: trastuzumab; Drug: paclitaxel; Drug: fluorouracil; Drug: epidoxorubicin; Drug: cyclophosphamide

INTERVENTIONS:
Drug: lapatinib — Arm B 1250mg/d PO Arm C 750mg/d PO
  Other Names: Tyverb/Tykerb
  Arms: Arm B; Arm C
Biological: trastuzumab — First dose 4mg/kg in 60mins, then weekly 2mg/kg in 30 mins
  Other Names: Herceptin
  Arms: Arm A; Arm C
Drug: paclitaxel — 80mg/sqm 1 hour infusion for 12 weeks
  Other Names: Taxol
Drug: fluorouracil — 600mg/sqm iv day 1 q21 days for four coursess
Drug: epidoxorubicin — 75mg/sqm iv day 1 q21 days for four courses
Drug: cyclophosphamide — 600mg/sqm day 1 q21 days for four courses

SUMMARY:
Evaluate the activity of Trastuzumab, Lapatinib, and a combination of both agents with chemotherapy in the preoperative (neoadjuvant) treatment of early breast cancer.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed infiltrating primary breast cancer of > 2.0 cm in largest clinical diameter

HER2 positive tumor (either IHC 3+ or FISH+)

* Availability of tumor tissue suitable for biological and molecular examination before starting primary treatment
* Age >18, < 65 years
* ECOG PS 0-1
* Normal organ and marrow function as defined below:

leukocytes ³ 3000/microL

absolute neutrophil count ³ 1,500/microL

platelets ³ 100,000/microL

total bilirubin <= 1.5x ULN. In case of Gilbert's syndrome, <2 x ULN is allowed

AST (SGOT)/ALT(SGPT)<= 2.5 X institutional upper limit of normal

Alkaline phosphatase <= 2.5 x ULN

Creatinine within normal institutional limits

* Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or MUGA scan
* Eligibility of patients receiving medications or substances known to affect, or with the potential to affect the activity or pharmacokinetics of lapatinib will be determined following review of their use by the Principal Investigator. A list of medications and substances known or with the potential to interact with CYP450 isoenzymes is provided
* The effects of lapatinib on the developing human fetus at the recommended therapeutic dose are unknown; women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately, the patient should be apprised of the potential hazard to the fetus and potential risk for loss of the pregnancy
* Ability to understand and the willingness to sign a written informed consent document
* Ability to swallow and retain oral medication

Exclusion criteria:

* Stage IIIB, IIIC, and inflammatory breast cancer
* Stage IV breast cancer
* Contraindication to the treatment with anthracycline, paclitaxel and/or trastuzumab
* Prior treatment with chemotherapy, endocrine therapy or radiotherapy. Prior treatment with EGFR targeting therapies
* Treatment with any other investigational agents, or with all herbal (alternative) medicines
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy or breastfeeding; (breast feeding should be discontinued to be enrolled in the study)
* Women of childbearing potential that refusal to adopt adequate contraceptive measures
* HIV-positive patients receiving combination anti-retroviral therapy
* GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)
* Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2006-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- GSK Investigational Site, Berlin, State of Berlin, Germany
- Italy (15):
  - GSK Investigational Site, Brindisi, Apulia
  - GSK Investigational Site, Carpi (MO), Emilia-Romagna
  - GSK Investigational Site, Forlì, Emilia-Romagna
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Piacenza, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Treviglio (BG), Lombardy
  - GSK Investigational Site, Candiolo (TO), Piedmont
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Cremona
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Perugia
  - GSK Investigational Site, Reggio Emilia
  - GSK Investigational Site, Varese
- GSK Investigational Site, Warsaw, Poland

REFERENCES:
- [Background] Guarneri V, Frassoldati A, Bottini A, Cagossi K, Bisagni G, Sarti S, Ravaioli A, Cavanna L, Giardina G, Musolino A, Untch M, Orlando L, Artioli F, Boni C, Generali DG, Serra P, Bagnalasta M, Marini L, Piacentini F, D'Amico R, Conte P. Preoperative chemotherapy plus trastuzumab, lapatinib, or both in human epidermal growth factor receptor 2-positive operable breast cancer: results of the randomized phase II CHER-LOB study. J Clin Oncol. 2012 Jun 1;30(16):1989-95. doi: 10.1200/JCO.2011.39.0823. Epub 2012 Apr 9. PMID 22493419
- [Derived] Guarneri V, Dieci MV, Griguolo G, Miglietta F, Girardi F, Bisagni G, Generali DG, Cagossi K, Sarti S, Frassoldati A, Gianni L, Cavanna L, Pinotti G, Musolino A, Piacentini F, Cinieri S, Prat A, Conte P; of the CHER-Lob study team. Trastuzumab-lapatinib as neoadjuvant therapy for HER2-positive early breast cancer: Survival analyses of the CHER-Lob trial. Eur J Cancer. 2021 Aug;153:133-141. doi: 10.1016/j.ejca.2021.05.018. Epub 2021 Jun 19. PMID 34153715
- [Derived] Guarneri V, Dieci MV, Frassoldati A, Maiorana A, Ficarra G, Bettelli S, Tagliafico E, Bicciato S, Generali DG, Cagossi K, Bisagni G, Sarti S, Musolino A, Ellis C, Crescenzo R, Conte P. Prospective Biomarker Analysis of the Randomized CHER-LOB Study Evaluating the Dual Anti-HER2 Treatment With Trastuzumab and Lapatinib Plus Chemotherapy as Neoadjuvant Therapy for HER2-Positive Breast Cancer. Oncologist. 2015 Sep;20(9):1001-10. doi: 10.1634/theoncologist.2015-0138. Epub 2015 Aug 5. PMID 26245675
- [Derived] Guarneri V, Generali DG, Frassoldati A, Artioli F, Boni C, Cavanna L, Tagliafico E, Maiorana A, Bottini A, Cagossi K, Bisagni G, Piacentini F, Ficarra G, Bettelli S, Roncaglia E, Nuzzo S, Swaby R, Ellis C, Holford C, Conte P. Double-blind, placebo-controlled, multicenter, randomized, phase IIb neoadjuvant study of letrozole-lapatinib in postmenopausal hormone receptor-positive, human epidermal growth factor receptor 2-negative, operable breast cancer. J Clin Oncol. 2014 Apr 1;32(10):1050-7. doi: 10.1200/JCO.2013.51.4737. Epub 2014 Mar 3. PMID 24590635

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants underwent core biopsy of the primary tumor, for the histological diagnosis and the biological characterization of the tumor. Radiological investigations were performed to rule out the metastatic disease. After diagnostic confirmation of the infiltrating carcinoma, participants were randomized to one of the three treatment arms.
Groups:
- Chemotherapy (CT) Plus Trastuzumab: Participants received chemotherapy (CT), which included paclitaxel 80 milligrams per meters squared (mg/m^2) weekly for 12 weeks, followed by intravenous (IV) fluorouracil 600 mg/m^2, IV epidoxorubicin 75 mg/m^2, and IV cyclophosphamide 600 mg/m^2, once every 21 days for four treatment courses. Trastuzumab was administered throughout the course of the CT and for two weeks after the last CT administration. The first dose of trastuzumab was administered at 4 milligrams per kilogram (mg/kg) IV for 60 minutes on the day of the first paclitaxel course. Subsequent administrations were given weekly at 2 mg/kg IV for 30 minutes. Treatments were administered for 26 weeks prior to surgery.
- CT Plus Lapatinib 1500 mg: Participants received CT, which included paclitaxel 80 mg/m^2 weekly for 12 weeks, followed by IV fluorouracil 600 mg/m^2, IV epidoxorubicin 75 mg/m^2, and IV cyclophosphamide 600 mg/m^2, once every 21 days for four treatment courses. Participants received lapatinib 1500 mg/day orally on an empty stomach throughout the course of the CT and for three weeks after the last CT administration. Treatments were administered for 26 weeks prior to surgery. Following Independent Data Monitoring Committee (IDMC) recommendations, lapatinib doses were reduced to 1250 mg/day orally on an empty stomach.
- CT Plus Trastuzumab and Lapatinib 1000 mg: Participants received CT, which included paclitaxel 80 mg/m^2 weekly for 12 weeks, followed by IV fluorouracil 600 mg/m^2, IV epidoxorubicin 75 mg/m^2, and IV cyclophosphamide 600 mg/m^2, once every 21 days for four treatment courses. Trastuzumab was administered throughout the course of the CT and for two weeks after the last CT administration. The first dose of trastuzumab was administered at 4 mg/kg IV for 60 minutes on the day of the first paclitaxel course. Subsequent administrations were given weekly at 2 mg/kg IV for 30 minutes. Participants received lapatinib 1000 mg/day orally on an empty stomach throughout the course of the CT and for three weeks after the last CT administration. Treatments were administered for 26 weeks prior to surgery. Following IDMC recommendations, lapatinib doses were reduced to 750 mg/day orally on an empty stomach.
Period: Overall Study
Arm/Group | Chemotherapy (CT) Plus Trastuzumab | CT Plus Lapatinib 1500 mg | CT Plus Trastuzumab and Lapatinib 1000 mg
Started | 36 | 39 | 46
Completed | 32 | 32 | 42
Not Completed | 4 | 7 | 4
Not completed — Disease Progression | 1 | 1 | 0
Not completed — Adverse Event | 2 | 5 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- CT Plus Trastuzumab: Participants received chemotherapy (CT), which included paclitaxel 80 milligrams per meters squared (mg/m^2) weekly for 12 weeks, followed by intravenous (IV) fluorouracil 600 mg/m^2, IV epidoxorubicin 75 mg/m^2, and IV cyclophosphamide 600 mg/m^2, once every 21 days for four treatment courses. Trastuzumab was administered throughout the course of the CT and for two weeks after the last CT administration. The first dose of trastuzumab was administered at 4 milligrams per kilogram (mg/kg) IV for 60 minutes on the day of the first paclitaxel course. Subsequent administrations were given weekly at 2 mg/kg IV for 30 minutes. Treatments were administered for 26 weeks prior to surgery.
- Total: Total of all reporting groups
Arm/Group | CT Plus Trastuzumab | CT Plus Lapatinib 1500 mg | CT Plus Trastuzumab and Lapatinib 1000 mg | Total
Number analyzed (Participants) | 36 | 39 | 46 | 121
Age, Continuous [Mean (Full Range); unit: Years] | 50 [34 to 65] | 49 [34 to 68] | 49 [26 to 65] | 49.3 [26 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 39 | 46 | 121
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 34 | 37 | 44 | 115
  Asian | 1 | 2 | 2 | 5
  Unknown | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathological Complete Response (pCR) in the Breast and in the Lymph Nodes
Description: Pathological Complete Response (pCR) is defined by the complete absence of infiltrating tumor cells in the breast and in the lymph nodes. The pathological response in the breast was evaluated according to the criteria of Miller and Payne as follows: Grade 1, no change or some alteration to individual malignant cells, but no reduction in overall cellularity; Grade 2, a minor loss in tumor cells (up to 30%); Grade 3, between an estimated 30% and 90% reduction in tumor cells; Grade 4, marked disappearance of tumor cells, with only a small cluster or a dispersed cell remaining (more than 90% loss); Grade 5, no identifiable malignant cells. Ductal carcinoma in situ (DCIS) may be present. Grades were interpreted as follows: Grade 1-2=no response; Grade 3-4=partial response; Grade 5=complete response. pCR was defined by comparing specimens obtained at Baseline (biopsy) to those obtained upon surgery.
Time Frame: At Baseline and surgery (within 5 weeks after the last chemotherapy administration) (assessed up to Study Week 29)
Population: Efficacy Analysis Population: all participants in the Intent-to-Treat Population (all participants who were randomized), except for the 2 participants who were excluded because of withdraw of consent and major protocol deviation
Measure: Number; unit: Percentage of participants
Arm/Group | CT Plus Trastuzumab | CT Plus Lapatinib 1500 mg | CT Plus Trastuzumab and Lapatinib 1000 mg
Number analyzed (Participants) | 36 | 38 | 45
Percentage of participants | 25 | 26.3 | 46.7
Statistical Analysis 1: Comparison: CT Plus Trastuzumab vs CT Plus Lapatinib 1500 mg vs CT Plus Trastuzumab and Lapatinib 1000 mg; Test type: Non-Inferiority or Equivalence — An exploratory comparison between the combined two single anti-HER2 arms and the dual anti-HER2 arm was performed (Arm 3 versus Arms 1 and 2); p = 0.019, Chi-squared — Exploratory analysis; percentage of participants = 25.0, 90% CI [13.1 to 36.9] — The estimated value represents the percentage of particpants in the CT plus trastuzumab treatment group with pathological complete response
Statistical Analysis 2: Comparison: CT Plus Lapatinib 1500 mg; Test type: Superiority or Other; percentage of participants = 26.3, 90% CI [14.5 to 38.1] — The estimated value represents the percentage of particpants in the CT plus lapatinib 1500 mg treatment group with pathological complete response
Statistical Analysis 3: Comparison: CT Plus Trastuzumab and Lapatinib 1000 mg; Test type: Superiority or Other; percentage of participants = 46.7, 90% CI 2-sided [34.4 to 58.9] — The estimated value represents the percentage of particpants in the CT plus traztuzumab plus lapatinib 1000 mg treatment group with pathological complete response

2. Secondary Outcome: Percentage of Participants With the Indicated Clinical Objective Response (Complete Response and Partial Response), Stable Disease, and Progressive Disease, as Assessed by Ultrasonography
Description: The clinical response was evaluated by comparing the tumor size (largest tumor diameter) before (at Baseline [biopsy]) and after treatment (before surgery), as assessed by ultrasonography examination. The clinical response was scored by Response Evaluation Criteria in Solid Tumors (RECIST) as follows: complete clinical response: the nodule is not detectable and all the ultrasound abnormality detected at diagnosis disappeared (margins circumscribed, round oval shape, parallel orientation, isoechoic echo pattern, no posterior acoustic features, echogenic lesion boundary, and tumor vascularity not present); partial clinical response: the longest diameter of the tumor has been reduced by >50%, and the ultrasound characteristics of the tumor persist; no response (stable disease): the longest diameter of the tumor has been reduced by <50% or has increased by no more than 20% from the starting value; progressive disease: tumor longest diameter has increased >20% from the starting value.
Time Frame: At Baseline and after primary treatment (within 2 weeks before surgery; up to Study Week 27)
Population: Efficacy Analysis Population
Measure: Number; unit: Percentage of participants
Arm/Group | CT Plus Trastuzumab | CT Plus Lapatinib 1500 mg | CT Plus Trastuzumab and Lapatinib 1000 mg
Number analyzed (Participants) | 36 | 38 | 45
Percentage of participants
  Complete Response (CR) | 30.5 | 15.8 | 42.2
  Partial Response (PR) | 41.7 | 44.7 | 28.9
  Stable Disease | 5.5 | 13.1 | 0
  Progressive Disease | 2.8 | 2.6 | 0
  Not Evaluable | 19.4 | 23.7 | 28.9

3. Secondary Outcome: Percentage of Participants Who Had Breast-conserving Surgery (BCS), Mastectomy, and Conversion From Mastectomy to BCS
Description: The percentage of participants who had BCS and mastectomy and who were initiallycandidates for mastectomy and who actually had BCS was measured. At Baseline, the surgeon stated, within 4 weeks before starting the primary treatment, which type of surgical treatment he would perform in the absence of primary therapy and in the case of primary therapy (if the tumor size was reduced by the primary treatment to less than 3 centimeters), and the reasons for these choices. The rules for choosing the type of surgical treatment are reported in the Consensus Conference on Primary Treatment of Early Breast Cancer. The surgeon was to have re-evaluated the participant after primary treatment. In cases in which the type of surgical procedure was different from that originally programmed, the reason for this chance was to have been reported.
Time Frame: At Baseline and at surgery (up to Study Week 29)
Population: Efficacy Analysis Population
Measure: Number; unit: Percentage of participants
Arm/Group | CT Plus Trastuzumab | CT Plus Lapatinib 1500 mg | CT Plus Trastuzumab and Lapatinib 1000 mg
Number analyzed (Participants) | 36 | 38 | 45
Percentage of participants
  BCS | 66.7 | 57.9 | 68.9
  Mastectomy | 33.3 | 39.5 | 31.1
  Conversion from mastectomy to BCS | 61.9 | 42.8 | 60

4. Secondary Outcome: Time to Treatment Failure From the Start of Primary Therapy
Description: Time to treatment failure (TTF) is defined as the interval of time between the date of randomization and the earliest date of disease progression, premature treatment discontinuation and death due to any cause. The overall disease progression date is the earlier of the two disease progression dates from ultrasonography and mammography assessments. For ultrasonography, disease progression is defined as at least 20% increase in the longest diameter of the primary lesion at pre-surgery comparing to Baseline. For mammography, disease progression is defined as at least 20% increase in the larger nodule dimension at pre-surgery comparing to Baseline. For participants who has neither progressed, pre-maturely withdrawn or died, time to treatment failure will be censored at the latest date of ultrasonography and mammography tumor assessments.
Time Frame: From randomization up to Study Week 307
Population: ITT Population: all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CT Plus Trastuzumab | CT Plus Lapatinib 1500 mg | CT Plus Trastuzumab and Lapatinib 1000 mg
Number analyzed (Participants) | 36 | 39 | 46
Months | 28.2 [28.2 to 59.8] | 39.6 [NA to NA] — The confidence limits for the median value are not estimable because there are no time points that satisfy the condition using the method of Klein and Moeschberger (1997). | 39.6 [6.3 to 39.6]

5. Secondary Outcome: Number of Participants With Treatment Failure
Description: Treatment failure is defined as the occurrence of local tumor progression (including ipsilateral and controlateral breast), distant tumor progression, permanent treatment discontinuation (either for the experimental or conventional arm), or death due to any cause.
Time Frame: From randomization up to 29 weeks
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | CT Plus Trastuzumab | CT Plus Lapatinib 1500 mg | CT Plus Trastuzumab and Lapatinib 1000 mg
Number analyzed (Participants) | 36 | 39 | 46
Participants | 7 | 9 | 7

6. Secondary Outcome: Percentage of Inhibition of Biomarkers Ki67, pAKT, pMAPK, Tunel Test, PTEN, and pEGFR After Treatment
Description: The percentage of inhibition of intermediate (EGFR, HER2, pMAPK, pAKT, PTEN, and PI3KCA) and final (TUNEL and Ki67) biomarkers of the proliferation and apoptosis pathways was calculated as the difference between the staining scores before (Baseline [biopsy]) and after treatment (withdrawal).
Time Frame: At Baseline and Withdrawal (assessed up to Study Week 29)
Population: ITT Population. Only those participants contributing data to the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of inhibition
Arm/Group | CT Plus Trastuzumab | CT Plus Lapatinib 1500 mg | CT Plus Trastuzumab and Lapatinib 1000 mg
Number analyzed (Participants) | 34 | 37 | 42
Percentage of inhibition
  Ki67, Baseline, n=34, 37, 42 | 25 [10 to 60] | 25 [4 to 70] | 30 [4 to 90]
  Ki67, Post-treatment, n=22, 21, 18 | 19 [1 to 50] | 15 [3 to 40] | 10 [1 to 30]
  pAKT, Baseline, n=34, 37, 42 | 2.5 [1 to 100] | 10 [0 to 90] | 0 [0 to 90]
  pAKT, Post-treatment, 18, 20, 17 | 0 [0 to 10] | 0 [0 to 90] | 0 [0 to 90]
  pMAPK, Baseline, n=9, 5, 7 | 0 [0 to 10] | 10 [0 to 80] | 0 [0 to 20]
  pMAPK, Post-treatment, n=0, 1, 2 | NA [NA to NA] — No participants were analyzed for pMAPK at this time point. | 70 [70 to 70] | 5 [0 to 10]
  Tunel test, Baseline, n=25, 27, 31 | 0.4 [0.05 to 2.6] | 0.58 [0.05 to 1.5] | 0.8 [0.05 to 2.5]
  Tunel test, Post-treatment, n=7, 12, 11 | 0.1 [0.05 to 1.1] | 0.1 [0.05 to 0.55] | 0.05 [0.05 to 0.4]
  PTEN, Baseline, n=27, 35, 37 | 80 [0 to 100] | 80 [0 to 100] | 90 [0 to 100]
  PTEN, Post-treatment, n=14, 17, 15 | 100 [10 to 100] | 80 [0 to 100] | 80 [0 to 100]
  pEGFR, Baseline, n=21, 24, 28 | 0 [0 to 80] | 0 [0 to 60] | 0 [0 to 70]
  pEGFR, Post-treatment, n=5, 10, 11 | 0 [0 to 90] | 0 [0 to 0] | 0 [0 to 5]

7. Secondary Outcome: Number of Participants With Any Adverse Event (AE), Including Serious Adverse Events (SAEs), Occurring in >=5% of Participants
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment had been exercised in deciding whether reporting was appropriate in other situations.
Time Frame: From the first dose of randomized therapy to 30 days after the last dose of randomized therapy (assessed up to Study Week 29)
Population: Safety Population: all randomized participants
Measure: Number; unit: Participants
Arm/Group | CT Plus Trastuzumab | CT Plus Lapatinib 1500 mg | CT Plus Trastuzumab and Lapatinib 1000 mg
Number analyzed (Participants) | 36 | 39 | 46
Participants | 35 | 38 | 46

8. Secondary Outcome: Number of Variations/Somatic Mutation in PI3KCA at Baseline
Description: Analysis of mutations in the PI3KCA gene was performed from RNA extracted from frozen tumor tissue samples (sections). A gene is either a wild-type (no mutation) or mutated (presence of a mutation). Exons 9 and 20 of the PI3KCA gene were accessed (high frequency mutation at these two spots).
Time Frame: Baseline
Population: ITT Population. Only those participants for which high-quality tumor tissue samples were available were analyzed.
Measure: Number; unit: Variations/Somatic mutations
Arm/Group | CT Plus Trastuzumab | CT Plus Lapatinib 1500 mg | CT Plus Trastuzumab and Lapatinib 1000 mg
Number analyzed (Participants) | 30 | 37 | 42
Variations/Somatic mutations
  PIK3CA Exon 9 Wild-Type | 29 | 35 | 39
  PIK3CA Exon 9 Mutation | 1 | 2 | 3
  PIK3CA Exon 20 Wild-type | 25 | 31 | 37
  PIK3CA Exon 20 Mutation | 5 | 6 | 5

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the first dose of randomized therapy to 30 days after the last dose of randomized therapy (up to Study Week 29).
Description: SAEs and non-serious AEs were collected for all participants who received at least one dose of study medication.
Arm/Group | CT Plus Trastuzumab | CT Plus Lapatinib 1500 mg | CT Plus Trastuzumab and Lapatinib 1000 mg
Serious Adverse Events (participants affected / at risk) | 14/36 | 13/39 | 21/46
Other Adverse Events (participants affected / at risk) | 35/36 | 38/39 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT Plus Trastuzumab (N=36) | CT Plus Lapatinib 1500 mg (N=39) | CT Plus Trastuzumab and Lapatinib 1000 mg (N=46)
Neutropenia (Blood and lymphatic system disorders) | 10 | 7 | 16
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 3
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Neutrophil count (Investigations) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Hyperpyrexia (General disorders) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT Plus Trastuzumab (N=36) | CT Plus Lapatinib 1500 mg (N=39) | CT Plus Trastuzumab and Lapatinib 1000 mg (N=46)
Diarrhoea (Gastrointestinal disorders) | 12 | 27 | 38
Nausea (Gastrointestinal disorders) | 22 | 18 | 26
Vomiting (Gastrointestinal disorders) | 13 | 16 | 22
Abdominal pain upper (Gastrointestinal disorders) | 4 | 10 | 12
Dyspepsia (Gastrointestinal disorders) | 5 | 8 | 10
Constipation (Gastrointestinal disorders) | 7 | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 5 | 6
Stomatitis (Gastrointestinal disorders) | 2 | 4 | 7
Haemorrhoids (Gastrointestinal disorders) | 1 | 2 | 9
Cheilitis (Gastrointestinal disorders) | 0 | 2 | 1
Lip dry (Gastrointestinal disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 22 | 19 | 31
Leukopenia (Blood and lymphatic system disorders) | 4 | 2 | 9
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 20 | 17
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 7 | 16
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 6 | 8
Erythema (Skin and subcutaneous tissue disorders) | 2 | 5 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 2 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 6
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 6
Acne (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Asthenia (General disorders) | 17 | 10 | 12
Pyrexia (General disorders) | 2 | 10 | 14
Fatigue (General disorders) | 7 | 6 | 6
Mucosal inflammation (General disorders) | 2 | 6 | 7
Oedema peripheral (General disorders) | 2 | 2 | 1
Influenza like illness (General disorders) | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 4 | 6 | 8
Aspartate aminotransferase increased (Investigations) | 1 | 5 | 4
Blood bilirubin increased (Investigations) | 0 | 2 | 3
White blood cell count decreased (Investigations) | 2 | 3 | 0
Ejection fraction decreased (Investigations) | 1 | 2 | 1
Haemoglobin decreased (Investigations) | 0 | 2 | 1
Neutrophil count decreased (Investigations) | 0 | 2 | 1
Headache (Nervous system disorders) | 6 | 5 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 5 | 8
Paraesthesia (Nervous system disorders) | 2 | 5 | 4
Syncope (Nervous system disorders) | 0 | 1 | 6
Dizziness (Nervous system disorders) | 2 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 2 | 1
Cystitis (Infections and infestations) | 3 | 2 | 6
Folliculitis (Infections and infestations) | 0 | 2 | 5
Pharyngitis (Infections and infestations) | 3 | 1 | 2
Conjunctivitis (Infections and infestations) | 1 | 2 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2 | 3
Influenza (Infections and infestations) | 1 | 0 | 3
Rhinitis (Infections and infestations) | 2 | 0 | 1
Hypertension (Vascular disorders) | 5 | 2 | 4
Hot flush (Vascular disorders) | 1 | 2 | 2
Hypotension (Vascular disorders) | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Drug hypersensitivity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4
Insomnia (Psychiatric disorders) | 4 | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 1 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 4
Dysuria (Renal and urinary disorders) | 0 | 2 | 4
Breast pain (Reproductive system and breast disorders) | 3 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.